CLINICAL TRIAL: NCT00066352
Title: A Phase II Study of PS-341 in Advanced or Metastatic Urothelial Cancer (Transitional Cell Cancer of the Bladder, Ureter, and Renal Pelvis)
Brief Title: Bortezomib in Treating Patients With Advanced or Metastatic Transitional Cell Cancer of the Bladder, Renal Pelvis, or Ureter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-018; CDR0000315537 (Registry Identifier: PDQ (Physician Data Query)); NCI-6150
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: recurrent bladder cancer; stage IV bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase II trial is studying how well bortezomib works in treating patients with advanced or metastatic transitional cell cancer of the bladder, renal pelvis, or ureter.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and duration of response in patients with advanced or metastatic transitional cell cancer of the bladder, renal pelvis, or ureter when treated with bortezomib.
* Determine the 1-year, median, and overall survival rate of patients treated with this drug.
* Determine the stable disease rate and duration and time to progression in patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Correlate baseline and post-treatment levels of NF-kappaB and HIF-1 alpha in tumor biopsies with clinical outcome in patients treated with this drug.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients in complete remission (CR) may receive up to 2 courses after confirmation of CR.

Patients are followed within 3 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study within approximately 6.6-17.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed transitional cell cancer of the urothelium, including the bladder, renal pelvis, or ureter

  * Advanced or metastatic disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1 OR
* Karnofsky 80-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST/ALT no greater than 3 times ULN (less than 5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 45 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able and willing to undergo biopsy of tumor lesions
* No other primary cancer requiring treatment within the past 3 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No grade 1 or greater peripheral neuropathy
* No ongoing or active infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 2 prior chemotherapy regimen for metastatic disease

  * Prior neoadjuvant or adjuvant therapy allowed provided it was completed more than 12 months prior to study entry
  * Patients who relapse within 12 months after completion of neoadjuvant or adjuvant therapy are allowed provided they did not receive chemotherapy for recurrent disease
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior chemotherapy as a radiosensitizer is allowed* NOTE: *May be administered concurrently with radiotherapy; may be in addition to a single line of therapy for locally advanced or metastatic disease

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* More than 4 weeks since prior myelotoxic radiotherapy (more than 3,000 cGy to fields including substantial bone marrow) and recovered
* No concurrent radiotherapy

Surgery

* At least 4 weeks since prior surgery for cancer of the urothelium (except nephrostomy tubes and ureteral stents)

Other

* At least 4 weeks since any prior therapy and recovered
* No other concurrent investigational or commercial agents or therapies intended to treat the malignancy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09; Primary Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Objective response by RECIST criteria every 6 weeks

SECONDARY OUTCOMES:
Objective response duration
Stable disease duration
Progression-free survival
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winquist, MD, Study Chair — London Health Sciences Centre
Locations (15):
- United States (11):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (4):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Gomez-Abuin G, Winquist E, Stadler WM, Pond G, Degendorfer P, Wright J, Moore MJ. A phase II study of PS-341 (Bortezomib) in advanced or metastatic urothelial cancer. A trial of the Princess Margaret Hospital and University of Chicago phase II consortia. Invest New Drugs. 2007 Apr;25(2):181-5. doi: 10.1007/s10637-006-9009-4. Epub 2006 Sep 16. PMID 16983508